CLINICAL TRIAL: NCT02983006
Title: A Phase 1 Study of TRAIL-DR5 Antibody DS-8273a Administered in Combination With Nivolumab in Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: Study of DS-8273a With Nivolumab in Unresectable Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Bristol-Myers Squibb (Industry); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00906
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Melanoma
Keywords: TRAIL-DR5; DS-8273a; Immunoglobulin gamma-1 (IgG1); Cell mediated cytotoxicity (ADCC); Complement dependent cytotoxicity (CDC); DR5; Immunoglobulin G4 (IgG4); Monoclonal antibody; Programmed Cell Death 1 (PD-1)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — DS-8273a; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DS-8273a & Nivolumab (Experimental): Patient groups (cohorts) will receive a single dose level of DS 8273a & Nivolumab; DS 8273a will be increased in subsequent cohorts.
  Interventions: Biological: DS-8273a; Biological: Nivolumab

INTERVENTIONS:
Biological: DS-8273a — * Starting Dose: 4 mg/ kg IVQ 3 weeks (Cohort 1)
  * Dose Escalation: 8 mg/kg IV Q 3 weeks (Cohort 2), 16 mg/kg IV Q 3 weeks (Cohort 3), 24 mg/kg IV Q 3 weeks (Cohort 4), 2 mg/kg IV Q 3 weeks (Cohort -1), 4 mg/kg IV Q 3 weeks (Cohort -2)
Biological: Nivolumab — 5 mg/kg IV Q 3 weeks
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, and immunoregulatory (pharmacodynamic; PD) activity of DS-8273a administered in combination with nivolumab (anti-PD-1 antibody) to subjects with unresectable Stage III or Stage IV melanoma.

DETAILED DESCRIPTION:
Principal investigator hypothesize that TRAIL D5 antibody DS-8273a administered in combination with nivolumab will be well tolerated and that the addition of DS-8273a will augment the clinical efficacy of nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* 1) Signed Written Informed Consent The signed informed consent form prior to the performance of any study related procedures that are not considered part of standard of care.

  2) Target Population
  1. Subjects who are ipilimumab naïve with progressive unresectable Stage III or Stage IV melanoma; eligible patients may have had prior adjuvant therapy, but not including ipilimumab, and been treated with up to 3 prior treatments for metastatic melanoma [eg, chemotherapy, other biologic or targeted therapy or Interleukin-2 (IL-2)].
  2. Histologic or cytologic confirmation of stage III or stage IV melanoma
  3. Measurable disease at baseline as assessed by CT and/or MRI
  4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
  5. Screening laboratory values must meet the following criteria and should be obtained within 7 days prior to registration • White blood cell (WBC) ≥ 2000/μL • Neutrophils ≥ 1500/μL

     * Platelets ≥ 100 x103/μL
     * Hemoglobin > 9.0 g/dL
     * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
     * Female CrCl = (140 - age in years) x weight in kg x 0.85
     * 72 x serum creatinine in mg/dL
     * Male CrCl = (140 - age in years) x weight in kg x 1.00
     * 72 x serum creatinine in mg/dL
     * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤ 3 x ULN Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

       3) Age and Reproductive Status Men and women ≥ 18 years old

  <!-- -->

  1. Men and women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study, and for women at least 23 weeks after the last dose of investigational product and for men at least 31 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. See Section 3.3.3 for the definition of WOCBP.
  2. Women must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.

     Exclusion Criteria:
* 1) Target Disease Exceptions

  a) Subjects with known or suspected brain metastasis, or brain as the only site of disease are excluded with the following exceptions.

  i) Subjects with controlled brain metastasis (no radiographic progression at least 4 weeks following radiation and/or surgical treatment, off steroids for at least 4 weeks, and have no new or progressing neurological signs or symptoms) will be allowed.

  b) Subjects with a history of prior malignancy with the exception of carcinoma in situ of the cervix or other malignancy diagnosed > 2 years ago that has undergone potentially curative therapy with no evidence of disease for the last ≥ 2 years and that is deemed by the investigator to be at a low risk of recurrence.

  2) Medical History and Concurrent Diseases

  a) Active autoimmune disease or a history of known or suspected autoimmune disease with the exception of subjects with isolated vitiligo, treated thyroiditis or resolved childhood asthma/atopy.

  b) Known human immunodeficiency virus (HIV), active hepatitis A, or hepatitis B or C infection.

  c) Evidence of active infection that requires anti-bacterial, anti-viral, or anti-fungal therapy ≤ 7 days prior to initiation of study drug therapy d) History of acute diverticulitis within the last 6 months, or current chronic diarrhea e) Active peptic ulcer disease even if asymptomatic f) Prior organ allograft or allogenic bone marrow transplantation g) Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following: i) Myocardial infarction within the past 6 months ii) Uncontrolled angina within the past 6 months iii) Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation or Torsades de pointes). Controlled atrial fibrillation by itself is not an exclusion criterion.

  h) Baseline toxicities from prior anti-cancer treatments > Grade 1. i) Inability to be venipunctured and/or tolerate venous access. j) Any major surgery within 4 weeks or a diagnostic procedure (eg incision, needle biopsy) within 1 day of study drug administration.

  k) Known drug or alcohol abuse. l) Presence of underlying medical condition that in the opinion of the Investigator or Sponsor could adversely affect the ability of the subject to comply with or tolerate study procedures and/or study therapy, or confound the ability to interpret the tolerability of combined administration of DS-8273A and nivolumab in treated subjects.

  3) Allergies and Adverse Drug Reaction

  a) History of allergy to components of nivolumab or DS-8273A, or known allergy to other antibody therapies.

  4) Sex and Reproductive Status
  1. WOCBP who are unwilling or unable to use an acceptable method to minimize the risk of pregnancy for the entire study period and for at least 23 weeks after the last dose of investigational product.
  2. Women who are pregnant or breastfeeding.
  3. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
  4. Sexually active fertile men not using effective birth control if their partners are WOCBP.

     5) Prohibited Prior Treatments and/or Therapies

  a) Exposure to any investigational drug within 4 weeks of study drug administration.

  b) Any anti-cancer therapy (eg, chemotherapy, biologics, radiotherapy, or hormonal treatment) within 4 weeks or at least 5 half-lives (whichever is longer) of study drug administration.

  c) Prior therapy with an anti-PD-1/PD-L1 antibody or a TRAIL-DR5 antibody d) Concurrent chemotherapy, hormonal therapy, immunotherapy regimens, or radiation therapy, standard or investigational.

  6) Other Exclusion Criteria
  1. Prisoners or subjects who are involuntarily incarcerated
  2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) of the protocol therapy | Up to 2 years
  Safety will be evaluated for all treated subjects using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Anti-tumor activity of the protocol therapy | Up to 2 years
  Tumor response will be determined for all subjects by RECIST 1.1 as well as by immune-related response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, MD, PhD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- Laura and Isaac Perlmutter Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Yoshida T, Ichikawa J, Giuroiu I, Laino AS, Hao Y, Krogsgaard M, Vassallo M, Woods DM, Stephen Hodi F, Weber J. C reactive protein impairs adaptive immunity in immune cells of patients with melanoma. J Immunother Cancer. 2020 Apr;8(1):e000234. doi: 10.1136/jitc-2019-000234. PMID 32303612